CLINICAL TRIAL: NCT03174925
Title: Elastography in Thyroid Nodule Evaluation
Brief Title: Ultrasound Elastography in Imaging Patients With Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aya Kamaya, Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-23634; NCI-2017-00841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); END0020 (Other: OnCore)
Record Dates: First submitted 2017-05-18; First posted 2017-06-05 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Malignant Thyroid Gland Neoplasm; Thyroid Gland Nodule
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Siemens Acuson S3000 ultrasound system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tissue Stiffness by Elastography (Experimental): Potentially cancerous thyroid nodules were assessed by elastrography, then a fine needle biopsy specimen or the surgically-excised nodule was assessed pathologically to determine cancer status.
  Interventions: Device: Siemens Acuson S3000 ultrasound system

INTERVENTIONS:
Device: Siemens Acuson S3000 ultrasound system — Shear Wave Elastography

SUMMARY:
This clinical trial studies how well ultrasound elastography works in assessing the cancer status of potentially malignant thyroid nodules.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Determine the utility of ultrasound elastography in evaluation of thyroid nodules being evaluated for the presence of cancer.

Elastography measures the passages of ultrasound shear waves through tissue to gauge the stiffness and compressibility of the tissue, collectively "tissue stiffness," and may be a better way to image thyroid nodules. Tissue stiffness is a physiological parameter that is being evaluated for differences between non-cancerous (benign) and cancerous thyroid nodules.

Participants will undergo elastography over the 10 minutes prior to either fine needle aspiration of a biopsy specimen or surgical resection of the thyroid nodule. Tissue specimens from the biopsy specimen or surgical resection will be assessed pathologically to determine actual cancer status.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a thyroid nodule that is amenable to ultrasound guided fine needle aspiration

Exclusion Criteria:

* Patients who are unable to lie supine for a biopsy
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tissue Stiffness by Elastography
Started | 55
Completed | 52
Not Completed | 3
Not completed — Elastographic images not retrievable | 2
Not completed — Elastography image not interpretable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tissue Stiffness by Elastography
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Stiffness of Thyroid Nodules as Measured by Elastography
Description: Potentially cancerous thyroid nodules will be assessed elastographically, and cancer status will be determined from a fine needle aspiration biopsy results or the surgically excised nodule. The outcome will be reported as median tissue stiffness with standard deviation for nodules that were determined non-cancerous (benign), cancerous, or indeterminate.
Time Frame: 1 week
Population: An individual participant could contribute multiple nodules.
Measure: Median (Standard Deviation); unit: meters/second
Units Other Than Participants: Thyroid nodules
Arm/Group | Tissue Stiffness by Elastography
Number analyzed (Participants) | 52
Number analyzed (Thyroid nodules) | 66
meters/second
  Pathologically Noncancerous Thyroid Nodules: number analyzed (Participants) | 35
  Pathologically Noncancerous Thyroid Nodules: number analyzed (Thyroid nodules) | 41
  Pathologically Noncancerous Thyroid Nodules | 2.7 (0.7)
  Pathologically Cancerous Thyroid Nodules: number analyzed (Participants) | 14
  Pathologically Cancerous Thyroid Nodules: number analyzed (Thyroid nodules) | 17
  Pathologically Cancerous Thyroid Nodules | 3.8 (0.7)
  Pathologically Indeterminate Thyroid Nodules: number analyzed (Participants) | 8
  Pathologically Indeterminate Thyroid Nodules: number analyzed (Thyroid nodules) | 8
  Pathologically Indeterminate Thyroid Nodules | 2.7 (1.1)

ADVERSE EVENTS:
Time Frame: Day of procedure
Arm/Group | Tissue Stiffness by Elastography
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT03174925/Prot_SAP_ICF_000.pdf